CLINICAL TRIAL: NCT05735366
Title: A Phase I Open-label, Multicenter Study to Evaluate the Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of SAIL66 in Patients With CLDN6-positive Locally Advanced or Metastatic Solid Tumors
Brief Title: A Phase 1 Study of SAIL66 in Patients With CLDN6-positive Locally Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SAL101JG
Record Dates: First submitted 2023-01-27; First posted 2023-02-21 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Q3W Dose Escalation part (Experimental): Patients will receive SAIL66 as tri-weekly IV infusions at escalated doses.
  Interventions: Drug: SAIL66
- Expansion part (Experimental): Patients will receive SAIL66 as a IV infusion at the recommended dose.
  Interventions: Drug: SAIL66
- QW Dose Escalation part (Experimental): Patients will receive SAIL66 as a weekly IV infusion at escalated doses.
  Interventions: Drug: SAIL66

INTERVENTIONS:
Drug: SAIL66 — SAIL66 as a IV infusion

SUMMARY:
This is a Phase 1 dose-escalation and expansion study that will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and preliminary efficacy of SAIL66 in patients with CLDN6-positive locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of signing Informed Consent Form
* Eastern Cooperative Oncology Group (ECOG) PS of 0 or 1
* Patient must have tumor specimen available for central pathology review and confirmed as CLDN6-positive
* (For male patients) Agreement to stay abstinent or use contraceptive measures with female partners, and agreement to refrain from donating sprerm during the treatment

Exclusion Criteria:

* Intending to become pregnant or breastfeed during the study and within 3 months after the last dose of SAIL66 or tocilizumab, whichever is longer
* Primary central nervous system (CNS) malignancy, symptomatic (seizures etc.) CNS metastases or CNS metastases required any anti-cancer treatment
* History or presence of CNS disease such as stroke (e.g., subarachnoid hemorrhage or cerebral infarction), epilepsy, CNS vasculitis, neurodegenerative disease, aphasia, dementia or paresis
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events of SAIL66[safety and tolerability] | From screening until study completion, treatment discontinuation or post-treatment follow up (approximately 18 weeks)
  Incidence, nature, and severity of adverse events graded according to NCI Common Terminology CTCAE v5.0, with severity of CRS determined according to the American Society for Transplantation and Cell Therapy (ASTCT) Consensus Grading Criteria
Change from baseline in vital signs[safety and tolerability] | From screening until study completion or treatment discontinuation (approximately 18 weeks)
  Change from baseline in vital signs
Change from baseline in clinical laboratory test results and examination findings[safety and tolerability] | From screening until study completion or treatment discontinuation (approximately 18 weeks)
  Change from baseline in clinical laboratory test results and examination findings specified in this study including, but not limited, electrocardiograms (ECGs)
Dose-limiting toxicities (DLTs) of SAIL66[safety and tolerability] | From Cycle 1 Day 1 until Cycle 1 Day 21 (Cycle 1 is 21 days)
  Incidence and nature of the DLTs [Q3W Dose Escalation part and QW Dose Escalation part]
Preliminary anti-tumor activity of SAIL66 when administered at selected dose(s) in each cohort [Expansion part] | From screening until study completion, treatment discontinuation or post-treatment follow up (approximately 18 weeks)
  Objective response rate (ORR), defined as the proportion of patients with a confirmed complete response (CR) or partial response (PR) on two consecutive occasions >= 4 weeks apart, assessed per Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 by the investigators.

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of SAIL66 [PK profile] | From screening until study completion, treatment discontinuation or post-treatment follow up (approximately 18 weeks)
  Maximum serum concentration (Cmax) of SAIL66
Trough serum concentration (Ctrough) of SAIL66 [PK profile] | From screening until study completion, treatment discontinuation or post-treatment follow up (approximately 18 weeks)
  Trough serum concentration (Ctrough) of SAIL66
Area under the concentration time-curve (AUC) of SAIL66 [PK profile] | From the first occurrence of CR or PR to progression disease (PD) or death from any cause (whichever occurs first) (approximately 18 weeks)
  Area under the concentration time-curve (AUC) of SAIL66
Objective response rate(ORR)[preliminary efficacy] | From screening until study completion, treatment discontinuation or post-treatment follow up (approximately 18 weeks)
  ORR assessed per RECIST v.1.1 by the investigators. [Q3W Dose Escalation part and QW Dose Escalation part]
Duration of response (DoR)[preliminary efficacy] | From the first occurrence of CR or PR to progression disease (PD) or death from any cause (whichever occurs first)(whichever occurs first) (approximately 18 weeks)
  Duration of response (DoR), defined as the time from the first occurrence of CR or PR to progression disease (PD) or death from any cause (whichever occurs first), per the investigator according to RECIST v.1.1
Disease control rate (DCR)[preliminary efficacy] | From screening until study completion, treatment discontinuation or post-treatment follow up (approximately 18 weeks)
  Disease control rate (DCR), defined as the proportion of patients who have CR, PR, or stable disease (SD) as best overall response per RECIST v.1.1 as determined by the investigator. SD must be confirmed at the first tumor assessment as scheduled in Appendix 1 after the start of treatment (the minimum duration for SD).
Progression-free survival (PFS)[preliminary efficacy] | From administration of first study treatment to the first occurrence of disease progression or death from any cause (approximately 18 weeks)
  Progression-free survival (PFS), defined as the time from administration of first study treatment to the first occurrence of disease progression or death from any cause, as determined by the investigator according to RECIST v.1.1
Overall survival (OS)[preliminary efficacy] | From administration of first study treatment to death from any cause (approximately 18 weeks)
  Overall survival (OS), defined as the time from administration of first study treatment to death from any cause [Expansion part]
Immunogenicity of SAIL66[preliminary efficacy] | From Cycle 1 Day 1 (Cycle 1 is 21 days) until study completion or treatment discontinuation (approximately 18 weeks)
  Incidence of ADAs to SAIL66 and potential correlation with PK parameters and safety

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Chugai Pharmaceutical Co. Ltd, Study Director — clinical-trials@chugai-pharm.co.jp
Locations (9):
- United States (5):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Japan (4):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Tokyo, Chuo Ku
  - Cancer Institute Hospital of JFCR, Tokyo, Koto Ku
  - Shizuoka Cancer Center, Shizuoka, Sunto-gun

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform. For further details on Chugai's Data Sharing Policy and how to request access to related clinical study documents, see here (www.chugai-pharm.co.jp/english/profile/rd/ctds_request.html).